CLINICAL TRIAL: NCT04872309
Title: MUlti-nuclear MR Imaging Investigation of Respiratory Disease-associated CHanges in Lung Physiology
Acronym: MURDOCH
Status: Suspended | Type: Observational
Why Stopped: COVID arm of study completed, paused while funding sought
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH20825
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Asthma; COPD; Covid19; Long COVID
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Asthma Patients: Adults with physician diagnosis of stable asthma (BTS guideline Step 3 or above).
- COPD Patients: Adults with Stage 3 or 4 COPD (as defined by GOLD guideline 2018)
- ICU COVID-19: Adults who have been hospitalised on ICU with COVID-19 (requiring CPAP or mechanical ventilation)
- Moderate/Severe COVID-19: Adults hospitalised with COVID-19
- Mild- Non-hospitalised COVID-19: Adult with proven COVID-19 infection, not hospitalised for COVID-19
- Non-hospitalised symptomatic (long-COVID group): Patients presenting at secondary care clinics post COVID-19 with ongoing symptoms.

SUMMARY:
Lung magnetic resonance imaging (MRI) with proton and inhaled inert gases has demonstrated a clinical ability to provide valuable structural and functional information in lung disease. Advances in lung MRI methods have led to the STH department handling clinical imaging referrals from local and national respiratory units. Hyperpolarised Xenon-129 gas MRI is now the gold-standard MRI modality used in clinical practice for asthma and COPD in Sheffield.

In this new study, the investigators will use Xenon gas MR imaging and 19F gas MR imaging to obtain physiological, structural, and functional information about patients with known respiratory disease, namely asthma and COPD. Up to 20 patients with asthma and up to 20 patients with COPD will be recruited. Study visits will involve lung function tests and imaging using proton MRI, hyperpolarised xenon gas MRI, and 19F perfluoropropane MRI. After initial baseline assessments, patients will be followed up after 3 and 6 years to investigate the utility of MRI and lung function measurements in tracking disease progression over time.

In addition, during the COVID-19 pandemic will also be studying the long term effects of this novel disease. The investigators will use Xenon gas MR imaging and pulmonary vascular 1H MR imaging to obtain physiological, structural, and functional information about patients with COVID-19, including hospitalised patients and mild, non-hospitalised COVID-19 patients. Participants may be invited for baseline assessments during the symptomatic phase of the disease and/or be followed up after 6, 12, 24 and 52 weeks (in line with clinical follow up for hospitalised patients) to investigate long term effects of this novel disease.

This novel approach will provide mechanistic insight in to clinical observations such as : (i) why previously healthy patients can respond so poorly to oxygen/ventilation therapy, (ii) why patients respond to proning, and (iii) whether this is caused by alveolar-capillary interstitial changes and /or microvascular clotting in the pulmonary vasculature (leading to V/Q mismatch), and (iv) whether these acute changes lead to long term interstitial lung disease.

DETAILED DESCRIPTION:
For asthma and COPD patients, this is a feasibility study to explore the use of gas MRI lung imaging techniques in tracking disease progression over a 6 year time period. Participants will have a baseline MRI scanning session and then be asked to come for repeat scans after 3 and 6 years.

Participants will attend for 3 visits, once at baseline, at 3years and 6 years. Each visit is split over 2 days should occur within one week. This is to ensure eligibility for MRI scanning.

At the eligibility visit the research team discuss study with patient and obtain informed consent. An MRI Screening Form is used to identify any contra-indications to MRI scanning. The participant will be asked further questions about their health, current diagnosis and any current treatments, smoking history, and about any exposure to pollutants either at home or at work. Women will be asked to take a urine pregnancy test, to ensure pregnant women are excluded from the study. The study doctor will perform a brief cardio-respiratory examination to check that it is safe for the patient to undertake the study. At the MRI scanning visit the participant will have a series of MRI scans, firstly using Xenon gas, then after a short break a they will have a second set of scans using 19F perfluoropropane gas. The participant will also undertake some simple lung function tests.

For COVID patients, this is pilot observational study using nationally unique MR imaging methods to investigate the acute and long-term pathophysiology of COVID-19 infection and the resulting changes seen in the lung, pulmonary vasculature and heart of patients with COVID-19 over the course of 12months.

Patients will attend for up to 5 visits. These are at baseline (patient may still be hospitalised, or this may be shortly after discharge) and 6, 12, 24 and 52 weeks post discharge. These visit timelines are designed to match with clinical follow up timelines for hospitalised patients. After the initial approach and consent patients will be screened for eligibility using the MRI scanning checklist. Patients who are still hospitalised or have significant ongoing respiratory problems will undertake a test gas inhalation under close supervision to ensure that this is tolerated prior to MRI scanning. A renal function blood test will be undertaken if required. For some non-hospitalised patients this will require an additional visit.

At the first MRI scanning visit consent will be taken or re-affirmed if taken prior to this visit. Medical history and medication check will be taken and women of child bearing age will undertake a pregancy test. The participant will have a series of MRI scans, firstly using Xenon gas, then after a short break a they will have a proton MRI which includes using gadolinium contrast. The participant will also undertake some simple lung function tests, including spirometry, gas transfer and endoPAT. Lung function tests will only be completed if the patient is non-infectious.

The repeat assessments at 6, 12, 24 and 52 weeks will be the same as the first visit, patients will be contacted prior to their repeat visit to repeat the MRI screening form and confirm eligibility.

ELIGIBILITY:
Asthma patients

Inclusion criteria

1. Adults aged 18 years or over.
2. Physician diagnosis of stable asthma (BTS guideline Step 3 or above).

Exclusion criteria

1. Recent asthma exacerbation requiring steroids and/or antibiotics in the 6 weeks prior to a study visit.
2. Asthma deemed by a physician to be unstable or in an active treatment modification phase.
3. Pregnancy (determined by urine pregnancy test for pre-menopausal women at the screening (V1) or eligibility visits (V3, V5).
4. Resting blood oxygen saturations (SaO2) < 90% in room air, as measured by oximeter.
5. Inability to comfortably lie supine.
6. Any contraindication(s) to MRI scanning as per the MRI Screening Form and standard operating procedure used by the Unit of Academic Radiology, Sheffield.
7. Disease or co-morbidity of sufficient severity as to make survival until 6 year follow up unlikely, as deemed by study clinician.

COPD patients

Inclusion criteria

1. Adults aged 18 years or over.
2. Stage 3 or stage 4 COPD as defined by GOLD guidelines 2018, (https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-v1.7-FINAL-14Nov2018-WMS.pdf) .
3. FEV1:FVC <0.7 (spirometry results).
4. FEV1 < 50% predicted (spirometry results). N.B. spirometry results that have been performed as part of a patient's normal clinical care within 6 months of study visit 1 may be used for definition of disease status and inclusion into the study; alternatively if no spirometry result is available it will be performed at visit 1.

Exclusion criteria

1. Recent COPD exacerbation requiring steroids and/or antibiotics in the 6 weeks prior to a study visit.
2. COPD deemed by a physician to be unstable or in an active treatment modification phase, including the active phase of pulmonary rehabilitation.
3. Pregnancy (determined by urine pregnancy test for pre-menopausal women at the screening (V1) or eligibility visits (V3, V5).
4. Significant heart failure as assessed by clinician.
5. Resting blood oxygen saturations (SaO2) < 90% in room air, as measured by oximeter.
6. Inability to comfortably lie supine.
7. Any contraindication(s) to MRI scanning as per the MRI questionnaire and standard operating procedure used by the Unit of Academic Radiology, Sheffield.
8. Disease or co-morbidity of sufficient severity as to make survival until 6 year follow up unlikely, as deemed by study clinician.

ICU COVID-19

Inclusion criteria

1. Adult over 18
2. Proven COVID-19
3. Hospitalised/previously hospitalised on ICU requiring CPAP or mechanical ventilation
4. Able to give informed consent
5. For currently hospitalised participants, or those with significant on-going respiratory problems - Tolerates test inhalation of non-polarised gas according to supervising clinicians' judgement AND SaO2 do not fall below 80%

Exclusion criteria

1. No previous diagnosed respiratory disease with the exception of mild asthma, defined as:

   1. no oral steroids in past year
   2. -no hospital admissions last year
   3. max 500mcg per day BDP or 250mcg fluticasone or equivalent ICS
2. Pregnancy (determined by urine pregnancy test for pre-menopausal women)
3. Significant heart failure as assessed by clinician.
4. Resting blood oxygen saturations (SaO2) < 90%, as measured by oximeter at the time of scanning.
5. Inability to comfortably lie supine.
6. Any contraindication(s) to MRI scanning or Gadolinium contrast agent as per the MRI questionnaire and standard operating procedure used by the MRI Unit.

6. Stage 4 or 5 chronic kidney disease, defined by creatinine clearance less than 30 mL/min as estimated by the Cockcroft-Gault equation (due to gadolinium contrast use). 7. Previous allergy to gadolinium contrast. 8. Significant co-morbidity to make enrolment unsuitable, as deemed by study clinician.

Moderate/Severe COVID-19

Inclusion criteria

1. Adult over 18
2. Proven COVID-19
3. Hospitalised/previously hospitalised with a diagnosis of pneumonia (chest X-ray or CT scan consistent with COVID-19 infection)
4. Whilst hospitalised had new onset oxygenation impairment defined as:

   a. An SpO2 ≤93% on room air and/or requiring additional oxygen to maintain satisfactory oxygenation
5. Able to give informed consent
6. For currently hospitalised participants, or those with significant on-going respiratory problems - Tolerates test inhalation of non-polarised gas according to supervising clinicians judgement AND SaO2 do not fall below 80%

Exclusion criteria

1. No previous diagnosed respiratory disease with the exception of mild asthma, defined as:

   1. no oral steroids in past year
   2. -no hospital admissions last year
   3. max 500mcg per day BDP or 250mcg fluticasone or equivalent ICS
2. Pregnancy (determined by urine pregnancy test for pre-menopausal women)
3. Significant heart failure as assessed by clinician.
4. Resting blood oxygen saturations (SaO2) < 90%, as measured by oximeter at time of MRI scanning.
5. Inability to comfortably lie supine.
6. Any contraindication(s) to MRI scanning or Gadolinium contrast agent as per the MRI questionnaire and standard operating procedure used by the MRI Unit.
7. Stage 4 or 5 chronic kidney disease, defined by creatinine clearance less than 30 mL/min as estimated by the Cockcroft-Gault equation (due to gadolinium contrast use).
8. Previous allergy to gadolinium contrast.
9. Significant co-morbidity to make enrolment unsuitable, as deemed by study clinician.

Mild- Non-hospitalised

Inclusion criteria

1. Adult over 18
2. Proven COVID-19
3. Not hospitalised for COVID-19
4. Able to give informed consent

Exclusion criteria

1. No previous diagnosed respiratory disease with the exception of mild asthma, defined as:

   1. no oral steroids in past year
   2. -no hospital admissions last year
   3. max 500mcg per day BDP or 250mcg fluticasone or equivalent ICS
2. Pregnancy (determined by urine pregnancy test for pre-menopausal women)
3. Significant heart failure as assessed by clinician.
4. Resting blood oxygen saturations (SaO2) < 90%, as measured by oximeter.
5. Inability to comfortably lie supine.
6. Any contraindication(s) to MRI scanning or Gadolinium contrast agent as per the MRI questionnaire and standard operating procedure used by the MRI Unit.
7. Stage 4 or 5 chronic kidney disease, defined by creatinine clearance less than 30 mL/min as estimated by the Cockcroft-Gault equation (due to gadolinium contrast use).
8. Previous allergy to gadolinium contrast.
9. Significant co-morbidity to make enrolment unsuitable, as deemed by study clinician.

Non-hospitalised symptomatic (long-COVID group)

Inclusion criteria

1. Adult over 18
2. Proven COVID-19
3. Not hospitalised for COVID-19
4. Able to give informed consent
5. Attended secondary care clinic with on-going symptoms.

Exclusion criteria

1. No previous diagnosed respiratory disease with the exception of mild asthma, defined as:

   1. no oral steroids in past year
   2. no hospital admissions last year
   3. max 500mcg per day BDP or 250mcg fluticasone or equivalent ICS
2. Pregnancy (determined by urine pregnancy test for pre-menopausal women)
3. Significant heart failure as assessed by clinician.
4. Resting blood oxygen saturations (SaO2) < 90%, as measured by oximeter at the time of scanning.
5. Inability to comfortably lie supine.
6. Any contraindication(s) to MRI scanning or Gadolinium contrast agent as per the MRI questionnaire and standard operating procedure used by the MRI Unit.
7. Stage 4 or 5 chronic kidney disease, defined by creatinine clearance less than 30 mL/min as estimated by the Cockcroft-Gault equation (due to gadolinium contrast use).
8. Previous allergy to gadolinium contrast.
9. Significant co-morbidity to make enrollment unsuitable, as deemed by study clinician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asthma/COPD/COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
%Ventilated volume | 3-6 years for asthma/COPD patients, 3-12months for COVID-19 participants
  a measurement derived from MRI images that quantifies the relative amount of lung that is ventilated, corrected for size.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Unit of Radiology, Univeristy of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided